CLINICAL TRIAL: NCT06006468
Title: Evaluating ImmuNe Changes in the Evolution of Pre Type 1 Diabetes With Adult Onset
Acronym: INCEPTiON
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: CRF525
Record Dates: First submitted 2023-06-20; First posted 2023-08-23 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes; Type 1 Diabetes Mellitus Maturity Onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Genetic risk of Type 1 diabetes: 750 individuals with the highest type 1 diabetes genetic risk
  Interventions: Genetic: High genetic risk for type 1 diabetes
- Genetic risk of coeliac disease: 750 individuals with the highest coeliac disease genetic risk
  Interventions: Genetic: High gentic risk for Coeliac disease
- Controls: 750 individuals with Neutral type 1 diabetes and coeliac disease genetic risk

INTERVENTIONS:
Genetic: High genetic risk for type 1 diabetes — in individuals without diabetes comparison of prevalence of islet auto antibodies between individuals at high genetic risk of type 1 diabetes versus controls
  Groups: Genetic risk of Type 1 diabetes
Genetic: High gentic risk for Coeliac disease — in individuals without Coeliac disease comparison of prevalence of anti tissue transglutaminase antibodies between individuals at high genetic risk of coeliac disease versus controls
  Groups: Genetic risk of coeliac disease

SUMMARY:
Little is known about how type 1 diabetes or coeliac disease develop in adults. Studies following children at risk of type 1 diabetes from birth have shown that the marker of type 1 diabetes autoimmunity (antibodies against the insulin producing cells in the pancreas (Glutamic Acid Decarboxylase Autoantibodies (GADA), Insulin Autoantibodies (IAA), Zinc Transporter 8 Autoantibodies (ZnT8), Anti-tyrosine phosphatase-like insulinoma antigen 2 (IA-2))) can develop many years before glucose levels are raised and diabetes is diagnosed. In adults, it is unclear when antibodies develop in relation to high blood glucose levels and the diagnosis of type 1 diabetes.

Similarly in coeliac disease it is unclear to what degree Tissue transglutaminase autoantibodies (TTG) in adults proceed the development of clinically diagnosed disease.

The investigators will use samples collected and stored in The Exeter 10,000 volunteer research bank (https://exetercrfnihr.org/about/exeter-10000/) and so no new sample collection is required. This includes ~8000 participants with no history of coeliac disease or diabetes at recruitment. The investigators wish to determine prevalence of autoantibodies in the background adult population split by the highest genetic risk for type 1 diabetes and separately coeliac disease compared to a control population with lower genetic risk for these conditions. The investigators will also evaluate the proportion of these identified cases progressing to clinically diagnosed disease.

The aim of this study is to investigate evidence of autoimmunity prior to disease development and generate pilot data for the validity of screening based on genetic predisposition for type 1 diabetes and coeliac disease.

DETAILED DESCRIPTION:
Detecting the early stages of type 1 diabetes in children is possible and has positive implications for clinical care.

Studies following children at risk of type 1 diabetes from birth have shown that islet autoantibodies against (Glutamic Acid Decarboxylase (GADA), Insulin (IAA), Zinc Transporter 8 (ZnT8), Anti-tyrosine phosphatase-like insulinoma antigen 2 (IA-2))) can develop many years before diabetes is diagnosed. This makes islet-autoantibodies an excellent biomarker of early disease with the development of multiple (≥2) positive islet-autoantibodies marking the first stage of type 1 diabetes. Many studies in children have looked at strategies for increasing islet autoantibody detection given the high numbers needed to test if screening at the whole population level. This includes targeting for autoantibody testing those with a type 1 diabetes: family history and/or raised genetic risk. Identifying type 1 diabetes early matters as it can reduce the proportion of cases presenting with severe symptoms including with diabetic ketoacidosis. This is coupled to recent FDA approval of Teplizumab therapy aiming to slow down the progression of early type 1 diabetes.

Little is known about the early development or early case detection of type 1 diabetes in adults despite representing the majority of all cases. Despite the potential benefits of pre-clinical type 1 diabetes detection in children very little is known about the stages of development of type 1 diabetes in adults. Therefore as noted in a recent Type 1 Diabetes research Steering Committee meeting "The optimal strategies for identification of at-risk adults needs to be studied". This is despite over half of all type 1 diabetes cases developing in adults. Our recent work examining adult-onset type 1 diabetes at presentation suggests that when adult-onset type 1 diabetes cases are defined robustly, characteristics include high type 1 diabetes genetic risk, rapid progression of C-peptide loss and high (>90%) rates of islet autoantibody positivity. Of these adult autoantibody positive cases ~60% were multi-autoantibody positive. Previous literature suggesting type 1 diabetes is a more benign disease in older adults likely reflects the increasingly recognised misclassification of clinically defined type 1 diabetes cases in this age group.

The high rates of islet autoantibodies at diagnosis and associated high genetic risk in adult-onset type 1 diabetes cases suggests targeted screening for early disease in this age group, using these biomarkers as undertaken in children, is a possibility. Studies recruiting first degree relatives of individuals have included adults (typically up to 45 years of age) showing detection of individuals at risk of type 1 diabetes is possible, even if progression from stage 1 to clinical disease appears reduced with increasing age at autoantibody detection. However, as in children, the majority of type 1 diabetes cases in adults develop in those without a family history of the disease and therefore genetic risk guided screening offers an attractive alternative strategy but research into the validity of this approach is lacking.

Little is known about early Coeliac disease development in adults. Coeliac disease is similarly increasingly recognised in adults but the early development of the disease is unclear. Development of coeliac disease is associated with raised genetic risk which can be captured by a coeliac genetic risk score. Recognition of coeliac disease is difficult particularly in adults and early detection has been suggested to be associated with improved outcomes.

Datasets with genetics and stored samples allow pragmatic insights into the feasibility of targeted screening for early adult-onset type 1 diabetes and coeliac disease.

The investigators will use samples collected and stored in The Exeter 10,000 adult volunteer research bank (https://exetercrfnihr.org/about/exeter-10000/) which includes ∼8000 participants with no history of diabetes at recruitment (a median 10 years ago (minimum 3 years since recruitment)). This will allow islet autoantibody measurement without the need for additional sample collection. All participants have genotype data available and have given permission for the Exeter 10,000 team to prospectively access their health records. This dataset allows a pragmatic and cost-effective assessment of using genetic predisposition to type 1 diabetes and coeliac disease to guide islet-autoantibody/ tissue-transglutaminase testing in adults. This will provide vital pilot data which can help guide future screening strategies for detecting pre-clinical type 1 diabetes and coeliac disease in adults.

ELIGIBILITY:
Inclusion Criteria:

* Exeter 10,000 study participants with stored serum samples
* Consent for samples & data to be used in further research.

Exclusion Criteria:

* Diagnosed with diabetes at time of original sample collection
* Diagnosed with coeliac disease at time of original sample collection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will use samples and data from the Exeter 10,000 cohort, a research bank of adult volunteers (https://exetercrfnihr.org/about/exeter-10000/). Stored serum samples are available (allowing islet autoantibody measurement) for all participants including ∼8000 participants with no history of diabetes at recruitment (a median 10 years ago (minimum 3 years since recruitment)). Additionally all participants have genotype data available and have given permission to the research team to prospectively access their health records.
Sampling Method: Probability Sample
Enrollment: 2250 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of multi-islet autoantibody positive participants | through sample analysis, approx 6 months
  ≥2 positive islet autoantibodies (GAD, IA-2, ZNT8, IAA) between genetic risk groups for type 1 diabetes

SECONDARY OUTCOMES:
Number of islet autoantibody positive participants | through sample analysis, approx 6 months
  ≥1 positive islet autoantibodies (GAD, IA-2, ZNT8, IAA) between genetic risk groups for type 1 diabetes
Number of multi-islet autoantibody positive participants developing Diabetes | through study follow up an average of 10 years
  number of cases developing type 1 diabetes
Number of participants with positive Tissue transglutaminase autoantibodies | through sample analysis, approx 6 months
  Number of positive Tissue transglutaminase autoantibody in genetic risk groups for coeliac disease
Number of participants developing Coeliac disease | through study follow up an average of 10 years
  number of cases developing Coeliac disease

CONTACTS AND LOCATIONS:
Overall Officials: Richard Oram, Dr, Principal Investigator — University of Exeter & Royal Devon University Healthcare NHS Foundation Trust
Locations (1):
- NIHR Exeter Clinical Research Facility (Royal Devon University Healthcare NHS Foundation Trust), Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Extend data available through external application process to university of Exeter

REFERENCES:
- [Background] Insel RA, Dunne JL, Atkinson MA, Chiang JL, Dabelea D, Gottlieb PA, Greenbaum CJ, Herold KC, Krischer JP, Lernmark A, Ratner RE, Rewers MJ, Schatz DA, Skyler JS, Sosenko JM, Ziegler AG. Staging presymptomatic type 1 diabetes: a scientific statement of JDRF, the Endocrine Society, and the American Diabetes Association. Diabetes Care. 2015 Oct;38(10):1964-74. doi: 10.2337/dc15-1419. PMID 26404926
- [Background] Ziegler AG, Rewers M, Simell O, Simell T, Lempainen J, Steck A, Winkler C, Ilonen J, Veijola R, Knip M, Bonifacio E, Eisenbarth GS. Seroconversion to multiple islet autoantibodies and risk of progression to diabetes in children. JAMA. 2013 Jun 19;309(23):2473-9. doi: 10.1001/jama.2013.6285. PMID 23780460
- [Background] Orban T, Sosenko JM, Cuthbertson D, Krischer JP, Skyler JS, Jackson R, Yu L, Palmer JP, Schatz D, Eisenbarth G; Diabetes Prevention Trial-Type 1 Study Group. Pancreatic islet autoantibodies as predictors of type 1 diabetes in the Diabetes Prevention Trial-Type 1. Diabetes Care. 2009 Dec;32(12):2269-74. doi: 10.2337/dc09-0934. Epub 2009 Sep 9. PMID 19741189
- [Background] Steck AK, Vehik K, Bonifacio E, Lernmark A, Ziegler AG, Hagopian WA, She J, Simell O, Akolkar B, Krischer J, Schatz D, Rewers MJ; TEDDY Study Group. Predictors of Progression From the Appearance of Islet Autoantibodies to Early Childhood Diabetes: The Environmental Determinants of Diabetes in the Young (TEDDY). Diabetes Care. 2015 May;38(5):808-13. doi: 10.2337/dc14-2426. Epub 2015 Feb 9. PMID 25665818
- [Background] Sims EK, Besser REJ, Dayan C, Geno Rasmussen C, Greenbaum C, Griffin KJ, Hagopian W, Knip M, Long AE, Martin F, Mathieu C, Rewers M, Steck AK, Wentworth JM, Rich SS, Kordonouri O, Ziegler AG, Herold KC; NIDDK Type 1 Diabetes TrialNet Study Group. Screening for Type 1 Diabetes in the General Population: A Status Report and Perspective. Diabetes. 2022 Apr 1;71(4):610-623. doi: 10.2337/dbi20-0054. PMID 35316839
- [Background] Ziegler AG, Kick K, Bonifacio E, Haupt F, Hippich M, Dunstheimer D, Lang M, Laub O, Warncke K, Lange K, Assfalg R, Jolink M, Winkler C, Achenbach P; Fr1da Study Group. Yield of a Public Health Screening of Children for Islet Autoantibodies in Bavaria, Germany. JAMA. 2020 Jan 28;323(4):339-351. doi: 10.1001/jama.2019.21565. PMID 31990315
- [Background] Mahon JL, Sosenko JM, Rafkin-Mervis L, Krause-Steinrauf H, Lachin JM, Thompson C, Bingley PJ, Bonifacio E, Palmer JP, Eisenbarth GS, Wolfsdorf J, Skyler JS; TrialNet Natural History Committee; Type 1 Diabetes TrialNet Study Group. The TrialNet Natural History Study of the Development of Type 1 Diabetes: objectives, design, and initial results. Pediatr Diabetes. 2009 Apr;10(2):97-104. doi: 10.1111/j.1399-5448.2008.00464.x. Epub 2008 Sep 24. PMID 18823409
- [Background] Ziegler AG, Hummel M, Schenker M, Bonifacio E. Autoantibody appearance and risk for development of childhood diabetes in offspring of parents with type 1 diabetes: the 2-year analysis of the German BABYDIAB Study. Diabetes. 1999 Mar;48(3):460-8. doi: 10.2337/diabetes.48.3.460. PMID 10078544
- [Background] Hagopian WA, Erlich H, Lernmark A, Rewers M, Ziegler AG, Simell O, Akolkar B, Vogt R Jr, Blair A, Ilonen J, Krischer J, She J; TEDDY Study Group. The Environmental Determinants of Diabetes in the Young (TEDDY): genetic criteria and international diabetes risk screening of 421 000 infants. Pediatr Diabetes. 2011 Dec;12(8):733-43. doi: 10.1111/j.1399-5448.2011.00774.x. Epub 2011 May 12. PMID 21564455
- [Background] Ziegler AG, Danne T, Dunger DB, Berner R, Puff R, Kiess W, Agiostratidou G, Todd JA, Bonifacio E. Primary prevention of beta-cell autoimmunity and type 1 diabetes - The Global Platform for the Prevention of Autoimmune Diabetes (GPPAD) perspectives. Mol Metab. 2016 Feb 22;5(4):255-262. doi: 10.1016/j.molmet.2016.02.003. eCollection 2016 Apr. PMID 27069865
- [Background] Winkler C, Schober E, Ziegler AG, Holl RW. Markedly reduced rate of diabetic ketoacidosis at onset of type 1 diabetes in relatives screened for islet autoantibodies. Pediatr Diabetes. 2012 Jun;13(4):308-13. doi: 10.1111/j.1399-5448.2011.00829.x. Epub 2011 Nov 8. PMID 22060727
- [Background] Herold KC, Bundy BN, Long SA, Bluestone JA, DiMeglio LA, Dufort MJ, Gitelman SE, Gottlieb PA, Krischer JP, Linsley PS, Marks JB, Moore W, Moran A, Rodriguez H, Russell WE, Schatz D, Skyler JS, Tsalikian E, Wherrett DK, Ziegler AG, Greenbaum CJ; Type 1 Diabetes TrialNet Study Group. An Anti-CD3 Antibody, Teplizumab, in Relatives at Risk for Type 1 Diabetes. N Engl J Med. 2019 Aug 15;381(7):603-613. doi: 10.1056/NEJMoa1902226. Epub 2019 Jun 9. PMID 31180194
- [Background] Thomas NJ, Jones SE, Weedon MN, Shields BM, Oram RA, Hattersley AT. Frequency and phenotype of type 1 diabetes in the first six decades of life: a cross-sectional, genetically stratified survival analysis from UK Biobank. Lancet Diabetes Endocrinol. 2018 Feb;6(2):122-129. doi: 10.1016/S2213-8587(17)30362-5. Epub 2017 Nov 30. PMID 29199115
- [Background] Diaz-Valencia PA, Bougneres P, Valleron AJ. Global epidemiology of type 1 diabetes in young adults and adults: a systematic review. BMC Public Health. 2015 Mar 17;15:255. doi: 10.1186/s12889-015-1591-y. PMID 25849566
- [Background] Harding JL, Wander PL, Zhang X, Li X, Karuranga S, Chen H, Sun H, Xie Y, Oram RA, Magliano DJ, Zhou Z, Jenkins AJ, Ma RCW. The Incidence of Adult-Onset Type 1 Diabetes: A Systematic Review From 32 Countries and Regions. Diabetes Care. 2022 Apr 1;45(4):994-1006. doi: 10.2337/dc21-1752. PMID 35349653
- [Background] Thomas NJ, Hill AV, Dayan CM, Oram RA, McDonald TJ, Shields BM, Jones AG; StartRight Study Group. Age of Diagnosis Does Not Alter the Presentation or Progression of Robustly Defined Adult-Onset Type 1 Diabetes. Diabetes Care. 2023 Jun 1;46(6):1156-1163. doi: 10.2337/dc22-2159. PMID 36802355
- [Background] Thomas NJ, Dennis JM, Sharp SA, Kaur A, Misra S, Walkey HC, Johnston DG, Oliver NS, Hagopian WA, Weedon MN, Patel KA, Oram RA. DR15-DQ6 remains dominantly protective against type 1 diabetes throughout the first five decades of life. Diabetologia. 2021 Oct;64(10):2258-2265. doi: 10.1007/s00125-021-05513-4. Epub 2021 Jul 16. PMID 34272580
- [Background] Thomas NJ, Walkey HC, Kaur A, Misra S, Oliver NS, Colclough K, Weedon MN, Johnston DG, Hattersley AT, Patel KA. The relationship between islet autoantibody status and the genetic risk of type 1 diabetes in adult-onset type 1 diabetes. Diabetologia. 2023 Feb;66(2):310-320. doi: 10.1007/s00125-022-05823-1. Epub 2022 Nov 10. PMID 36355183
- [Background] Eason RJ, Thomas NJ, Hill AV, Knight BA, Carr A, Hattersley AT, McDonald TJ, Shields BM, Jones AG; StartRight Study Group. Routine Islet Autoantibody Testing in Clinically Diagnosed Adult-Onset Type 1 Diabetes Can Help Identify Misclassification and the Possibility of Successful Insulin Cessation. Diabetes Care. 2022 Dec 1;45(12):2844-2851. doi: 10.2337/dc22-0623. PMID 36205650
- [Background] Foteinopoulou E, Clarke CAL, Pattenden RJ, Ritchie SA, McMurray EM, Reynolds RM, Arunagirinathan G, Gibb FW, McKnight JA, Strachan MWJ. Impact of routine clinic measurement of serum C-peptide in people with a clinician-diagnosis of type 1 diabetes. Diabet Med. 2021 Jul;38(7):e14449. doi: 10.1111/dme.14449. Epub 2020 Nov 22. PMID 33131101
- [Background] Munoz C, Floreen A, Garey C, Karlya T, Jelley D, Alonso GT, McAuliffe-Fogarty A. Misdiagnosis and Diabetic Ketoacidosis at Diagnosis of Type 1 Diabetes: Patient and Caregiver Perspectives. Clin Diabetes. 2019 Jul;37(3):276-281. doi: 10.2337/cd18-0088. PMID 31371859
- [Background] Thomas NJ, Lynam AL, Hill AV, Weedon MN, Shields BM, Oram RA, McDonald TJ, Hattersley AT, Jones AG. Type 1 diabetes defined by severe insulin deficiency occurs after 30 years of age and is commonly treated as type 2 diabetes. Diabetologia. 2019 Jul;62(7):1167-1172. doi: 10.1007/s00125-019-4863-8. Epub 2019 Apr 10. PMID 30969375
- [Background] Jacobsen LM, Bocchino L, Evans-Molina C, DiMeglio L, Goland R, Wilson DM, Atkinson MA, Aye T, Russell WE, Wentworth JM, Boulware D, Geyer S, Sosenko JM. The risk of progression to type 1 diabetes is highly variable in individuals with multiple autoantibodies following screening. Diabetologia. 2020 Mar;63(3):588-596. doi: 10.1007/s00125-019-05047-w. Epub 2019 Nov 25. PMID 31768570
- [Background] Karges B, Prinz N, Placzek K, Datz N, Papsch M, Strier U, Agena D, Bonfig W, Kentrup H, Holl RW. A Comparison of Familial and Sporadic Type 1 Diabetes Among Young Patients. Diabetes Care. 2021 May;44(5):1116-1124. doi: 10.2337/dc20-1829. Epub 2021 Apr 6. PMID 33824143
- [Background] Cappello M, Morreale GC, Licata A. Elderly Onset Celiac Disease: A Narrative Review. Clin Med Insights Gastroenterol. 2016 Jul 27;9:41-9. doi: 10.4137/CGast.S38454. eCollection 2016. PMID 27486350
- [Background] Sharp SA, Jones SE, Kimmitt RA, Weedon MN, Halpin AM, Wood AR, Beaumont RN, King S, van Heel DA, Campbell PM, Hagopian WA, Turner JM, Oram RA. A single nucleotide polymorphism genetic risk score to aid diagnosis of coeliac disease: a pilot study in clinical care. Aliment Pharmacol Ther. 2020 Oct;52(7):1165-1173. doi: 10.1111/apt.15826. Epub 2020 Aug 13. PMID 32790217
- [Background] Corrao G, Corazza GR, Bagnardi V, Brusco G, Ciacci C, Cottone M, Sategna Guidetti C, Usai P, Cesari P, Pelli MA, Loperfido S, Volta U, Calabro A, Certo M; Club del Tenue Study Group. Mortality in patients with coeliac disease and their relatives: a cohort study. Lancet. 2001 Aug 4;358(9279):356-61. doi: 10.1016/s0140-6736(01)05554-4. PMID 11502314
- [Background] Aboulaghras S, Piancatelli D, Taghzouti K, Balahbib A, Alshahrani MM, Al Awadh AA, Goh KW, Ming LC, Bouyahya A, Oumhani K. Meta-Analysis and Systematic Review of HLA DQ2/DQ8 in Adults with Celiac Disease. Int J Mol Sci. 2023 Jan 7;24(2):1188. doi: 10.3390/ijms24021188. PMID 36674702